CLINICAL TRIAL: NCT07278297
Title: Parkinson Ballroom Fitness: The Impact of Personalized Dance on Motor- and Nonmotor Symptoms in People With Parkinson's
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1-10-72-46-25
Record Dates: First submitted 2025-11-21; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease (PD); Exercise Training; Dance Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-Fit group (Experimental)
  Interventions: Other: PB-Fit intervention
- Waitlist-control group (Other): This group will contribute as a control group as the PB-Fit group undergo the 7-week intervention. After the post assessment this group will also the receive the 7-week intervention.
  Interventions: Other: PB-Fit intervention

INTERVENTIONS:
Other: PB-Fit intervention — The intervention is 7 weeks of Parkinson Ballroom Fitness. A dance exercise program made specifically for persons with Parkinson Disease. This the first study to assess the effects of Parkinson Ballroom Fitness on motor and non-motor symptoms in persons with Parkinson Disease.

SUMMARY:
Parkinson Ballroom-Fitness (PB-Fit) is a group-based dance program developed for people with Parkinson's disease. Through music and movement at three different levels (seated, standing, and walking), participants work on balance, gait, strength, and coordination, while also experiencing joy, social connection, and renewed vitality.

The purpose of the present research project is to investigate whether seven weeks of PB-Fit training can improve gait and balance and enhance well-being and quality of life, and whether any effects are maintained twelve weeks after the intervention ends. The study is a randomized controlled trial with approximately forty participants and is conducted in collaboration with the Danish Parkinson's Association.

The PB-Fit program is based on dance styles such as waltz, swing, and Latin, and is individually adapted. Training takes place in small groups, where participants learn basic steps and work with both motor and cognitive challenges. The program is evidence-informed but lacks quantitative evaluation, which is the aim of this study.

PB-Fit is more than training-it is a community rooted in music, smiles, and meaningful relationships, where people with Parkinson's disease, regardless of functional level, are given the opportunity to experience joy, strength, and hope. This was clearly illustrated in the TV2 documentary "As Long as We Dance," in which several participants on the trip to Mallorca described their enthusiasm and the meaningfulness of PB-Fit.

The study is led by Associate Professor Martin Langeskov Christensen, PhD (Regional Hospital Viborg), in collaboration with Aarhus University and dance instructor Elisabeth Dalsgaard. The results will be published in an international scientific journal and shared with both professionals and participants.

Support from the Jascha Foundation will enable the study to be carried out and provide people with Parkinson's disease access to a meaningful, joyful, and evidence-based form of exercise. The long-term goal is to expand PB-Fit nationally and establish it as a permanent training option within municipalities and patient organizations across the country.

DETAILED DESCRIPTION:
Protocol Version 2, 23.04.2025

Parkinson Ballroom Fitness: The impact of personalized dance on motor- and nonmotor symptoms in people with Parkinson's

Members of the study group:

Principal Investigator:

Martin Langeskov Christensen, Associate Professor, PhD, Dept. of Clinical Medicine, Aarhus University and Researcher at Dept. of Neurology, Viborg Regional Hospital.

Co-investigators:

Theo S. Christensen, Scientific Assistant, MSc, Neurology, Viborg Regional Hospital.

Lars G. Hvid, Associate Professor, PhD, Aarhus University and Senior Researcher at The Danish MS Hospitals in Ry and Haslev.

Elisabeth Dalsgaard, Dance instructor and exercise physiologist, Owner of Swingtime Aps.

Background

Parkinson's disease (PD) is a chronic neurodegenerative disorder of the central nervous system characterized by the progressive loss of dopaminergic neurons in the substantia nigra. This loss leads to the cardinal motor symptoms of PD, including bradykinesia, rigidity, tremor, and postural instability . These motor symptoms significantly impair balance and walking capacity in individuals with PD, contributing to decreased quality of life and increased risk of falls .1 Moreover, problems with walking, balance and falls become increasingly important to people with PD as the condition progresses.2

Walking capacity in people with PD can be assessed through various tests, including the six spot step test (SSST) that involves challenging components of coordination and dynamic balance3, the Timed Up and Go (TUG) test as a measure of functional mobility, and falls risk prediction4, as well as 'fast' and 'endurance' walk tests such as the 10-meter walk test (10MWT)5 and the 6-minute walk test (6MWT)6, respectively . Balance impairments can be comprehensively assessed using tools such as the mini Balance Evaluation Systems Test (mini-BESTest), which evaluates dynamic balance, functional mobility, and gait .7-9 Additionally, The (modified) Four Square Step Test (mFSST10 / FSST11) can evaluate dynamic standing balance while stepping in multiple directions, and can be completed while requiring little equipment, space, and time in multiple rehabilitation settings. Furthermore, patient-reported outcomes such as the Parkinson's Disease Questionnaire (PDQ-39) can provide insights into the impact of PD on daily life and well-being12-14, whereas the Generic walking scale (Walk-12G)15,16 assesses the patient-reported impact of PD on different aspects of walking ability.

Exercise interventions, including those involving dance, have been shown effective in improving motor function and quality of life in people with PD.17 Interestingly, dance-based exercise appears particularly potent in terms of targeting impairments in balance, gait, and coordination through rhythmic and repetitive movements, offering both physical and cognitive benefits .18,19 However, more research is needed to determine its effects on non-motor symptoms and quality of life (QOL).19,20 Moreover, many dance modalities exist and ballroom dancing has received very little attention in this context21,22 with no evidence regarding the effectiveness of personalized dance interventions tailored to the functional levels and needs of individuals with PD.

Dance instructor and exercise physiologist Elisabeth Dalsgaard has developed a dance-based concept entitled Parkinson Ballroom Fitness (PB-Fit), specifically adapted for individuals with PD. This program focuses on the joy of movement and inclusion, with three difficulty levels corresponding to different overall disability categories (sitting, standing, and walking). Of note, the Danish Parkinson's Association previously received support to implement the project "Dance with Parkinsons". In the period 2017 to 2019, this project enabled the training of PB-Fit dance instructors and contributed to facilitating dance lessons for people with PD and their relatives all over Denmark. Yet this dance-based concept still awaits scientific evaluation in relation to motor and non-motor symptoms and QoL.

Study aims

Consequently, the main purpose of this study is to examine whether 7 weeks of PB-Fit (group-based personalized dance program) can improve walking capacity (primary outcome: SSST) and balance, alongside mental well-being and QoL in individuals with PD. An additional purpose is to evaluate these outcomes after 12 weeks of follow-up to determine the maintenance of potential dance-induced improvements and any behavioral changes. Of note, patients sitting in a wheelchair will also be included, but data from these participants will be analyzed separately in a secondary analysis.

Study hypothesis

We hypothesize that:

7 weeks of PB-Fit will elicit substantial improvements in walking capacity (particularly as measured by the SSST) and balance.

These improvements will be associated with enhancements in well-being and quality of life.

These improvements can be partly maintained after 12 weeks of follow-up, mainly due to behavioral changes such as participants continuing to dance.

Methods

Study design and inclusion criteria

A 7-week single-blinded, randomized controlled trial (RCT) will be conducted (Figure 1). Participants with PD will be recruited through social media platforms and local branches of the Danish Parkinson's Association. Clusters of participants (n=8-15) will be randomized to either the PB-Fit group or a waitlist control group when an adequate number has been identified and enrolled at one local branch/site. Baseline testing will precede randomization, and both groups will be re-evaluated post-interventions and the initial PB-Fit group again after a 12-week follow-up period.

The waitlist control group will continue their habitual lifestyle during the 7-week intervention period yet receive the same PB-Fit intervention afterwards.

Inclusion criteria:

Age ≥ 40 years

Clinical PD diagnosis

Ability to attend testing and dancing classes independently or with a caregiver / family

Exclusion criteria:

Comorbidities that prevent participation in the intervention

Moderate to severe cognitive impairment (Montreal Cognitive Assessment Test (MoCA) <18)

Recent fractures or critical physical impairments

Participation in structured exercise therapy (including dancing) in the past 3 months (≥ 2 sessions per week of moderate-to-high intensity)

The assessor will be blinded to the intervention arms at baseline, post, and follow-up. The study will be carried out following the regulations of the local scientific ethics committee and the Helsinki Declaration. All subjects will be informed about the purpose and the benefits/risks related to the study and have to provide written informed consent to participate.

PB-Fit Intervention

The intervention consists of 7 weeks of group-based PB-Fit sessions (2 per week). Group sizes will be approx. n=8-15 participants. The program, specifically adapted to PD, includes various dances (e.g., Latin, Waltz, Swing, HipHop) with different tempos to accommodate varying abilities. The concept is based on learning basic steps across the different dances, irrespective of disability level (sitting, standing, walking). Different tempos are presented, thereby enabling the participants to choose the rhythm according to their own starting point. Whilst the dances may differ in terms of taxing different bodily/physiological/functional aspects, these are the main aspects that are being targeted:

Balance: Each dance step is a weight transfer - and thus balance training.

Muscle strength: Involvement of both the lower and upper body hold aspects of muscle strength training.

Coordination: Steps and arms must be coordinated both in single steps and in small series.

Gait function: Gait is improved by training steps and following a certain rhythm.

Attitude. Continued training of the posture, especially from the standard dances, is evident. The dance invites you to focus on the attitude.

Fitness/endurance: Regardless of whether it is the fast or slow dances, it involves fitness/endurance training.

Of note, in sitting people with PD there is a predominant focus on coordination of the arms and cognitive skills, on strength in the arms and possibly in the legs, and on movement of the legs.

Progression of the PB-Fit will be done by increasing the duration of the sessions (from 40 minutes in week 1-2, to 60 minutes in week 6-7), the number of repetitions and minutes performing each dance exercise (from 3 x 2-3 minutes in week 1-2, to 4 x 5-6 minutes in week 6-7), and the complexity of tasks.

Outcome Measures

All outcome measures will be assessed at baseline (0 weeks), post (7 weeks), and follow-up (19 weeks). Patients in wheelchairs will only perform the walking and balance tests if considered feasible.

Primary outcome:

The six spot step test (SSST)3,23-25

Secondary outcomes:

Balance: miniBEST 26, the tandem test (part of the short physical performance battery (SPPB))

Walking capacity: Timed up and go (TUG, traditional and dual task version)27, 10MWT5, the 6-minute walk test (6MWT)6, Generic walking scale (Walk-12G)15,16

Mental well-being: WHO five well-being index (WHO-5) 28

Quality of life: the Parkinson's Disease Questionnaire (PDQ-39)12-14

Fatigue: Modified Fatigue Impact Scale (MFIS)29,30, Parkinson Fatigue Scale (PFS)31

Fall risk: Falls Efficacy Scale-International (FES-I)32

Physical activity: Baecke Physical Activity Questionnaire33

Non-motor symptoms: Non-Motor Symptoms Questionnaire (NMSQ)34

Trunk impairments: Trunk Impairment Scale 2.0 (TIS2)35,36

Sleep quality: Pittsburgh Sleep Quality Index (PSQI)37

Freezing of gait: New Freezing of Gait Questionnaire (NFOGQ)38

Adherence: The Exercise Adherence Rating Scale (EARS)39

Pain: King's Parkinson's Pain Questionnaire40

Cognitive function: Montreal Cognitive Assessment Test (MoCA)41, Executive function.

Statistical considerations

The study will be powered based on the primary outcome measure SSST, relying on data from a previous study in people with PD3,25. A mean SSST score of 8.1±1.8 seconds was used for the control group. A change of ±2.2 seconds in this test has been shown to reflect a true change surpassing measurement error in people with PD25, and a similar change (i.e., ≥2.1) has been found clinically important on a group level in multiple sclerosis patients.42 A two-sample two-sided power calculation showed a total of n=20 participants should be enrolled in each group (α = 0.01; power = 0.9; control mean post intervention 8.1±1.8 seconds; PB-Fit mean post intervention 5.9±1.8 seconds; dropout rate = 25%). Incorporating a 25% dropout rate, a total of n=50 people with PD will be enrolled, as a minimum, in the present study. This calculation includes only participants who are able to walk. In addition, a separate group of wheelchair users, expected to include approximately 10 participants, will be enrolled beyond the calculated total for the primary outcome. If there is a greater demand for participation in the study than our sample size calculation shows, we will include them accordingly.

Research plan

The described project is planned to be carried out by a scientific assistant from September 2025 until September 2026, under the supervision of Associate Professor, PhD, Martin Langeskov Christensen (primary investigator). The scientific assistant will work closely with a project manager from the Danish Parkinson's Association (Parkinsonforeningen), who will manage and organize participant inclusion and communication. Physiotherapy or sports science student assistants will carry out the testing, whereas dance instructors that have undertaken the official PB-Fit course (Parkinson Ballroom Fitness™) will carry out the intervention / dance lessons.

Plan for dissemination

The project's results will result in at least one scientific article to be published in a peer-reviewed international scientific journal (e.g., Movement Disorders). Results will be published whether positive, negative, or inconclusive. In addition, we will contribute to the knowledge sharing at the international research front by attending conferences (e.g., World Parkinson Congress). The acquired knowledge will be communicated to the involved participants, but also more broadly through the Danish Parkinson's Association.

Side effects and risks

PB-Fit can lead to muscle soreness, fatigue, joint pain, and dizziness due to the physical activity involved. The primary risks include falls and injuries from balance and coordination issues, overexertion, and mental fatigue from learning new steps. These factors will be considered for the safety and well-being of the participants. There are no other noticeable side effects or risks by participating in the outlined project.

Benefits and perspectives

Documenting and understanding the benefits of PB-Fit is of high relevance to patients with PD (and other chronic neurological conditions). First, the PB-Fit can be specifically tailored to the disability level (i.e., relating to the sitting, standing, walking categories) of any participant, and can therefore be carried out in groups that embrace the diversity of being a PD patient. Few (if any) other exercise concepts are designed this way. Second, the present study can help reveal whether task-specific training (in this case the task of doing complex and demanding balance/body control activities) can elicit positive adaptations across different aspects of balance and body control. Third, the proposed exercise modality (PB-Fit) is inexpensive, can be carried out in groups, and can be carried out in proximity of the homes of participants. Altogether, if the proposed PB-Fit study turns out to be effective (e.g., by improving both balance and well-being), we will have the evidence to support nationwide use of this concept. This will not only have benefits from an individual perspective, but also from a societal perspective (i.e., any attempt to postpone disability progression will likely reduce disability-related costs).

Ethics statement

The methods described in the project do not raise any special ethical concerns, and participation in the trial is considered to be close to risk-free for the participants involved. Additionally, the project will be registered at all relevant authorities (The Regional Committees on Health Research Ethics for Central Denmark Region; ClinicalTrials.gov). Subjects can leave the project at any time without any consequences. Results from the project will be published whether positive, negative or inconclusive.

Data management

The project complies with the legislation on the processing of personal data, i.e., the General Data Protection Regulation and the Danish Data Protection Act. The project will be registered at The Regional Committees on Health Research Ethics for Central Denmark Region. Data security and control are further ensured and overlooked by the Data-management group at Regional Hospital Central Jutland. Data is processed within Regional Hospital Central Jutland and all information and data collected will be treated confidentially by the personnel associated with the project. Of note, no data will be obtained from patient journals.

Economy

The project is initiated by the project responsible Associate Professor Martin Langeskov Christensen (Regional Hospital Central Jutland) together with Associate Professor Lars Hvid (Aarhus University) and Dance instructor Elisabeth Dalsgaard (Swingtime Aps). We will apply for funding to help cover the salary of dance instructors and test personnel as well as running costs (e.g., travel for project responsible) all which will be administered by Regional Hospital Central Jutland.

Compensation

Participants will not receive any compensation for travel costs associated with the test and training days.

Recruitment of participants and informed consent form

All participants will be recruited through the Danish Parkinson's Association. Specifically, a notice will be posted on their website and as a supplement to the inclusion of potential participants, an e-mail will be sent to the relevant local branches of the Danish Parkinson's Association, which can notify their members about the project via e-mail/newsletter. With approval of the various local branches of the Danish Parkinson's Association, the same information is potentially published/posted by the various local branches (primarily Facebook). If the project responsible or project employee are contacted by interested participants, they will receive the written material about the project, and asked for permission to be contacted by phone after 7 days or more by the project responsible or project employee. If the participants agree to be contacted, an exact date for an undisturbed information conversation (physical meeting or video meeting) will be scheduled, also emphasizing the possibility of participation of a support person (family member, friend etc.). During the private and undisturbed conversation it will be stated that (1) it is a request for participation in a health science research project, (2) the participants will be informed about the project's aims, benefits as well as risks and side effects, and (3) the written patient information will be reviewed. The leaflet "Før du beslutter dig" will also be given to the patient. There will also be time for questions. If the patient is still interested in participating (up to one week's reflection time is given), written informed consent will be given at the first physical meeting between the project responsible or project employee.

Patients Compensation Association

The Danish Patient Compensation Association covers participants in the project.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Clinical PD diagnosis
* Ability to attend testing and dancing classes independently or with a caregiver / family

Exclusion Criteria:

* Comorbidities that prevent participation in the intervention
* Moderate to severe cognitive impairment (Montreal Cognitive Assessment Test (MoCA) <18)
* Recent fractures or critical physical impairments
* Participation in structured exercise therapy (including dancing) in the past 3 months (≥ 2 sessions per week of moderate-to-high intensity)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Six Spot Step Test (SSST) | 25 weeks (from baseline assessment to post assessment = 7 weeks + 12 weeks follow-up period)

CONTACTS AND LOCATIONS:
Locations (1):
- Viborg Regional Hospital, Viborg, Central Jutland, Denmark